CLINICAL TRIAL: NCT01055912
Title: Multicenter, Randomized, Double-Blind, Placebo- Controlled, Parallel Group, Efficacy and Safety Study to Evaluate the Effects of Oral Administration of Lixivaptan in Patients With Congestive Heart Failure
Brief Title: Study to Evaluate the Effects of Oral Administration of Lixivaptan in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry)
Responsible Party: Cesare Orlandi, MD, SVP, Clinical Development, Cardiokine Bioharma, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CK-LX2401
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-11

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Volume Overload
MeSH Terms: conditions — Heart Failure; Edema | interventions — lixivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixivaptan (Experimental): Capsule, 100mg Lixivaptan or matching placebo once daily.
  Interventions: Drug: Lixivaptan
- Placebo (Placebo Comparator): Patients will be screened for entry into the study and will be randomized (2:1) to lixivaptan or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lixivaptan — Capsule. Patients will be screened for entry into the study and will be randomized (2:1) to lixivaptan or placebo. One hundred (100) patients will be randomized to receive lixivaptan 100 mg once daily (QD) for 8 weeks. Fifty (50) placebo patients will receive matching oral placebo for 8 weeks.
  Arms: Lixivaptan
Drug: Placebo — Patients will be screened for entry into the study and will be randomized (2:1) to lixivaptan or placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of oral lixivaptan capsules in patients with congestive heart failure.

DETAILED DESCRIPTION:
Diuretics are used extensively in the treatment of patients with CHF, and their efficacy is well established. However, there is a tendency for currently used diuretics to increase afterload and deplete electrolytes, and in many patients ventricular function continues to deteriorate over time.

Loop diuretics, such as furosemide, also have known negative effects on renal function reducing the glomerular filtration rate, and have been shown to activate the RAA system.

Lixivaptan is a potent, non-peptide selective antagonist of the vasopressin V2 receptor.

Lixivaptan treatment results in increased free water excretion, thus decreasing urine osmolality, increasing urine flow, and increasing serum osmolality. Short-term treatment with lixivaptan has demonstrated improved fluid management and electrolyte balance in HF patients.

This study was designed to assess the effects of vasopressin blockade with lixivaptan in patients with CHF with volume overload. A placebo-control arm will allow for assessment of the effect of lixivaptan in addition to standard diuretic therapy as compared with standard diuretic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and to provide signed and dated informed consent.
* Men and women aged 18 years or older.
* History of chronic CHF defined as requiring standard HF treatment (including diuretics) for a minimum of 30 days.
* Documented LVEF by any method within 12 months prior to screening.
* The patient has clinical evidence of volume overload at the time of inclusion with at least one of the following:

  * Dyspnea
  * Pulmonary congestion (rales)
  * Peripheral edema
  * Increased jugular venous pressure and/or hepatic congestion with ascites
  * Chest x-ray consistent with CHF
  * Plasma brain natriuretic peptide (BNP) ≥150 pg/mL or N-terminal prohormone brain natriuretic peptide (NT pro-BNP) ≥450 pg/mL

Exclusion Criteria:

* Women who are pregnant (positive pregnancy test), breastfeeding, or who will not adhere to the reproductive precautions as outlined in this protocol and in the informed consent form (ICF).
* Sustained (three blood pressure measurements over 1 hour) systolic blood pressure <90 mmHg at Screening or Day 0.
* ST segment elevation myocardial infarction or stroke within 30 days prior to Screening.
* Hemodynamically destabilizing cardiac arrhythmia within 30 days prior to Day 0.
* Clinically significant valvular disease.
* Known clinically significant obstructive, restrictive, or hypertrophic cardiomyopathy.
* Cardiac surgery or percutaneous coronary intervention within 30 days prior to Day 0.
* Major surgical procedure within 7 days prior to Day 0.
* Likely to undergo cardiac transplantation, left ventricular assist device (LVAD) or other device implantation, or other cardiac surgery within 3 months after Screening.
* Placement of implantable cardioverter defibrillator or cardiac resynchronization therapy device within 60 days prior to Day 0.
* CHF due to uncorrected thyroid disease, active myocarditis, or known amyloid cardiomyopathy.
* Presence of any clinically significant (as determined by the Investigator) endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, oncologic, and/or other major disease that might interfere with safe and compliant participation in this study.
* Screening laboratory findings as follows:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal
  * Total bilirubin >2.0 mg/dL
  * Serum creatinine >3.0 mg/dL
  * Hemoglobin <9.0 g/dL
* Uncontrolled diabetes mellitus as defined by the Investigator (e.g., glycosylated hemoglobin [HbA1c] >9%).
* History of chronic drug/medication abuse within the past 6 months; or current alcohol abuse.
* Co-morbid condition with an expected survival of less than 3 months.
* Known allergy to any vasopressin antagonist or any condition for which treatment with a vasopressin antagonist may present undue risk to the patient.
* Current or recent administration (within 7 days of Day 0) of prohibited medications as listed in Section 8.6.4 .
* Participation in any other investigational study of drugs or devices within 30 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of lixivaptan treatment in congestive heart failure (CHF) patients with volume expansion. | 8 weeks

SECONDARY OUTCOMES:
To assess the effects of lixivaptan treatment in CHF patients with volume expansion. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Phoenix Clinical, Phoenix, Arizona
  - Nea Clinic, Jonesboro, Arkansas
  - Capitol Interventional Cardiology, Carmichael, California
  - Merced Heart Associates, Merced, California
  - Orange County Heart Institute and Research Center, Orange, California
  - Innovative Research of West Florida, Inc, Clearwater, Florida
  - Edgewater Medical Research Inc, Edgewater, Florida
  - Foundation/Research/Cardiovascular Specialists Lower Keys, Key West, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Tampa Clinical Research, Tampa, Florida
  - Executive Health and Research Associates, Inc, Atlanta, Georgia
  - In-Quest Medical Research, LLC, Duluth, Georgia
  - Fox Valley Clinical Research Center, Aurora, Illinois
  - Maine Research Associates, Auburn, Maine
  - Primary Care Cardiology Research, Inc, Ayer, Massachusetts
  - Horizon Research, St Louis, Missouri
  - Great Lakes Medical Research, Westfield, New York
  - Raleigh Cardiology, Raleigh, North Carolina
  - Clinical Research Limited, Canton, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - East Texas Cardiology, Houston, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Ghali JK, Orlandi C, Abraham WT; CK-LX2401 Study Investigators. The efficacy and safety of lixivaptan in outpatients with heart failure and volume overload: results of a multicentre, randomized, double-blind, placebo-controlled, parallel-group study. Eur J Heart Fail. 2012 Jun;14(6):642-51. doi: 10.1093/eurjhf/hfs051. Epub 2012 Apr 17. PMID 22510424